CLINICAL TRIAL: NCT01427439
Title: A Prospective Epidemiological Research on Functioning Outcomes Related to Major Depressive Disorder
Acronym: PERFORM
Status: Completed | Type: Observational
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 13504A
Record Dates: First submitted 2011-08-26; First posted 2011-09-01 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Non-interventional study; Observational study
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Major Depressive Disorder

SUMMARY:
The purpose of this study is to describe patient functioning and examine associations between depressive symptoms and measures of the various roles of functioning.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a current or new diagnosis of major depressive episode (MDE) according to the Diagnostic and Statistical Manual of Mental Disorders IV Text Revision (DSM-IV-TR); diagnosis will be confirmed through the Mini International Psychiatric Interview (MINI) questionnaire (depression module)
* Outpatients starting an antidepressant treatment in monotherapy at baseline (treatment initiation or first treatment switch) as decided by the treating physician
* The patient will present within the normal course of care, for either a first or subsequent episode of depression

Exclusion Criteria:

* Schizophrenia or other psychotic disorders
* Bipolar disorder
* Dementia or other neurodegenerative disease significantly impacting cognitive functioning
* Mood disorder due to a general medical condition or substances
* Acute suicidality
* Patient treated for depression by a combination of different antidepressant treatments at the time of the consultation

Other exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from outpatient clinics (General Practitioner (GP) or psychiatrist)
Sampling Method: Non-Probability Sample
Enrollment: 1455 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Patients' functioning assessed by the Sheehan Disability Scale (SDS) total score | At baseline
Patients' functioning assessed by the SDS total score | At 12 months

SECONDARY OUTCOMES:
Associations between the patients' clinical condition measured as score on Clinical Global Improvement Severity scale (CGI-S) and of patients' functioning measured as total score on SDS | At baseline
Associations between the patients' clinical condition measured as score on CGI-S and of patients' functioning measured as total score on SDS | At 12 months
Associations between the patients' clinical condition measured as score on CGI-S and of patients' functioning measured as total score on SDS | At 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- FR, Paris, France

REFERENCES:
- [Derived] Haro JM, Hammer-Helmich L, Saragoussi D, Ettrup A, Larsen KG. Patient-reported depression severity and cognitive symptoms as determinants of functioning in patients with major depressive disorder: a secondary analysis of the 2-year prospective PERFORM study. Neuropsychiatr Dis Treat. 2019 Aug 13;15:2313-2323. doi: 10.2147/NDT.S206825. eCollection 2019. PMID 31616147
- [Derived] Haro JM, Lamy FX, Jonsson B, Knapp M, Brignone M, Caillou H, Chalem Y, Hammer-Helmich L, Rive B, Saragoussi D. Characteristics of patients with depression initiating or switching antidepressant treatment: baseline analyses of the PERFORM cohort study. BMC Psychiatry. 2018 Mar 27;18(1):80. doi: 10.1186/s12888-018-1657-3. PMID 29587672